CLINICAL TRIAL: NCT03155984
Title: Establishing Monitoring Strategies in Individuals With Prior Hepatitis B Virus Exposure Undergoing Anti-CD20 Antibody Containing Chemotherapy: A Prospective Observational Study
Brief Title: Optimizing HBV Management During Anti-CD20 Antibodies
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wai-Kay Seto, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW15-384
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Liver Dysfunction; Immune Suppression; Hepatitis B
MeSH Terms: conditions — Liver Diseases; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anti-CD20 antibody: Patients with hematological malignancies receiving anti-CD20 antibody therapy
  Interventions: Drug: Anti-CD20 antibody

INTERVENTIONS:
Drug: Anti-CD20 antibody — All patients receiving anti-CD20 therapy (rituximab, ofanumumab, obinutuzumab) for hematological malignancies

SUMMARY:
Hepatitis B virus (HBV) reactivation is common during anti-CD20 containing chemotherapy, even in HBsAg-negative patients with only prior HBV exposure. The optimal timing of commencing antiviral therapy and the interval of clinical monitoring is uncertain. 25% of the Hong Kong population has prior HBV exposure. The investigators plan monitor this cohort of patients and determine (1) the optimal time point for starting antiviral therapy based on the progression of HBV reactivation, and (2) the optimal interval of clinical monitoring.

DETAILED DESCRIPTION:
The use of immunosuppressive cytotoxic therapy in patients with chronic hepatitis B virus (HBV) infection is known to be associated with potentially fatal HBV reactivation. Prophylactic nucleoside analogue therapy has been shown to reduce the rates of HBV reactivation in hepatitis B surface antigen (HBsAg)-positive subjects, and is now recommended in current treatment guidelines.

Patients who are negative for HBsAg and anti-HBsAg antibody (anti-HBs) may be naïve to HBV. Nonetheless in HBV-endemic regions, such patients might have been infected with HBV and achieved HBsAg seroclearance. Prior HBV exposure is evidenced by the presence of positive antibody to the hepatitis B core antigen (anti-HBc). Hence although a HBsAg-negative, anti-HBc positive state may represent resolved HBV infection, it could also represent occult HBV infection with HBV persisting at low replicative levels following HBsAg seroclearance. Reactivation of HBV is then possible.

Rituximab, ofanumumab and obinutuzumab are chimeric monoclonal antibodies against the B-cell surface antigen CD20, and are used extensively in B-cell lymphoid malignancies and many non-malignant immune-mediated diseases in the fields of rheumatology, dermatology, neurology and nephrology.Previous retrospective and prospective studies have found the rates of HBV reactivation in HBsAg-negative, anti-HBc positive individuals who undergo anti-CD20 antibody containing chemotherapy to vary between 8.9 and 23.8%. This variation can be partially explained by the use of different definitions of HBV reactivation, including a combination of biochemical hepatitis, HBsAg seroreversion, or HBV DNA levels over a certain threshold. Another important factor was the lack of regular monitoring following commencement of anti-CD20 antibodies. In view of these discrepancies, our research team conducted a prospective study in which HBsAg-negative, anti-HBc positive lymphoma patients were monitored at 4-week intervals for up to 2 years following commencement of rituximab. Using a detectable serum HBV DNA level as the definition of HBV reactivation, the 2-year cumulative reactivation rate was 41.5%. Anti-HBs negativity was significantly associated with a higher risk of HBV reactivation.

Despite previous accurate description of the rate of HBV reactivation, many clinical questions remain :

1. Which is the better strategy for HBsAg-negative, anti-HBc positive patients receiving anti-CD20 antibodies - prophylactic antiviral therapy for all patients, or regular clinical monitoring and prescription of antiviral therapy when needed? Although prophylactic antiviral therapy has been proven effective, one needs to consider the high seroprevalence of anti-HBc in the HBV-endemic regions of East Asia that could reach 40%. Based on our two studies of rituximab and hematopoietic stem cell transplantation, the seroprevalence of anti-HBc in Hong Kong was between 26.4 and 27.6%. Universal prescription of antiviral therapy for all HBsAg-negative, anti-HBc positive individuals might not be cost-effective. At the same time, a recent technical review by the American Gastroenterological Association stated that based on current evidence, they "had no comment" on whether routine clinical monitoring could substitute prophylactic antiviral therapy.
2. If routine clinical monitoring were chosen, what is the optimal interval of monitoring? A current recommendation of every 1-3 months was based on expert opinion only. To answer this question, a prospective study is needed to observe the serial changes in HBV DNA levels over time in patients following the development of detectable HBV DNA, with each time epoch assessed for its suitability in monitoring.
3. Are all HBV reactivations clinically relevant? Our previous study only provided the rate of HBV DNA detectability, and did not describe its subsequent clinical progression. Will patients continue to have serial increases in HBV DNA level leading to biochemical hepatitis and/or HBsAg seroreversion, or do HBV DNA levels remain relatively low? A recent study found discrepancies between the rates of HBsAg seroconversion and HBV DNA ≥2,000 IU/mL (10.3% and 17.9% respectively), implying not all patients with HBV DNA detectability proceed to a progressive increase in HBV DNA levels, HBsAg seroreversion or biochemical hepatitis. Serial prospective data on this with respect to the cyclical treatment regimen of anti-CD20 antibodies are lacking.

The investigators propose a prospective observational study to answer these clinical questions and provide a concise management strategy for the large number of patients prescribed anti-CD20 antibodies containing therapy for both malignant and non-malignant diseases

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance score of ≤2.
3. HBsAg-negative, anti-HBc positive patient receiving anti-CD20 containing chemotherapy with or without antibody to the hepatitis B surface antigen (anti-HBs).
4. Baseline normal serum alanine amiontransferase (ALT) (≤30 U/L for men, ≤19 U/L for women).

Exclusion Criteria:

1. Concomitant liver diseases including chronic hepatitis C and D infection, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis.
2. Significant alcohol intake (>30 grams per day).
3. History of prior anti-HBV therapy, hematopoietic stem-cell transplantation, anti-CD20 antibody therapy, anti-CD52 antibody therapy or anti-tumour necrosis factor antibody therapy.
4. Baseline detectable HBV DNA (≥10 IU/mL). These patients will be started on prophylactic entecavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBsAg-negative anti-HBc positive individuals with hematological malignancies undergoing anti-CD20 containing chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
HBV Reactivation | From commencement of anti-CD20 antibody therapy for up to 2 years
  HBV DNA >= 10 IU/mL

SECONDARY OUTCOMES:
HBV-related hepatitis | From commencement of anti-CD20 antibody therapy for up to 2 years
  ALT >60 U/L for men; >38 U/L for women; and HBV DNA >2,000 IU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Kay Seto, MD, Principal Investigator — wkseto@hku.hk
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No such plan